CLINICAL TRIAL: NCT05174728
Title: Innovations in Placental Metabolism and Association With Antioxidants and Nutrients in Diabetes and Gestational Obesity
Acronym: IMPACTING
Status: Suspended | Type: Observational
Why Stopped: COVID-19 Pandemic
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); University of Cambridge (Other); Université Montpellier (Other); Universidade Federal do Rio de Janeiro (Other); Maternidade Escola da UFRJ (Unknown)
Responsible Party: Principal Investigator, Tatiana El Bacha Porto, Principal Investigator, Rio de Janeiro State University
Other Study IDs: 66949217.0.0000.5275
Record Dates: First submitted 2021-11-04; First posted 2022-01-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy Complications; Obesity, Maternal; Diabetes Mel Gestational - in Pregnancy
Keywords: pregnancy; gestational diabetes mellitus; pre-gestational maternal obesity
MeSH Terms: conditions — Pregnancy Complications; Pregnancy in Obesity; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, placental tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research project aims to investigate, in an innovative way, the molecular pathophysiology of gestational complications induced by maternal obesity and gestational diabetes mellitus (GDM). These complications have an immediate impact on obstetric outcomes - such as pre-eclampsia and intrauterine growth restriction - as well as long-term consequences for the health of the mother and child. This proposal aims to advance the understanding of the relationship between subclinical maternal and placental inflammation with dietary components through a prospective cohort of pregnant women. To this end, a prospective cohort of pregnant women will be conducted with four follow-up waves: 13th-20th (baseline), 24th-28th, 32nd-36th gestational weeks and at the time of delivery. Retrospective data referring to the first trimester of pregnancy will be obtained from the medical records. Pregnant women will be invited to participate in the study by registering at the prenatal service. Women who start prenatal care with less than 13 weeks of gestation will be registered, for capture in the 2nd consultation. The initial sample calculation is 120 volunteers. Maternal blood samples will be collected at 2 times: 2nd trimester appointment and 3rd trimester appointment. Placental and umbilical cord blood samples will be collected immediately after delivery. Dietary consumption during pregnancy will be assessed by 2 24-hour recalls at each visit (1 in person and 1 by telephone). The identification of functional biomarkers in maternal blood and placenta will serve for prognostic purposes of gestational complications such as Gestational Diabetes Mellitus. The identification of dietary factors associated with obesity and gestational diabetes mellitus and associated complications will provide information that will serve as a basis for nutritional guidelines for pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years;
* Free from chronic non-communicable diseases such as high blood pressure and type 2 diabetes mellitus, except obesity;
* Free from infectious diseases;
* Carrying a single fetus;
* Intention to deliver at Maternity School-Federal University of Rio de Janeiro

Exclusion Criteria:

* Smokers;
* With low weight in early pregnancy (BMI < 18.5 kg/m²). They will be verified by interview, before the signing the informed consent form.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of pregnant women with a single fetus, aged between 18-45 years who attended prenatal care at the Maternity School at Federal University of Rio de Janeiro. The study group includes healthy pregnant women, pregnant women with obesity and gestational diabetes mellitus associated or not with obesity.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Maternal redox homeostasis | between 24th and 28th gestational week
  Redox homeostasis will be assessed in maternal blood using a biological assay to measure the capacity of the sample to prevent the oxidation of a known fluorescence probe, in the presence of an oxidant. The unit of measure is concentration of plasma expressed as equivalent to a know antioxidant (after performing a calibration curve).
Maternal redox homeostasis [change] | between 34th and 35th gestational week
  Redox homeostasis will be assessed in maternal blood using a biological assay to measure the capacity of the sample to prevent the oxidation of a known fluorescence probe, in the presence of an oxidant. The unit of measure is concentration of plasma expressed as equivalent to a know antioxidant (after performing a calibration curve).
Fetal (cord blood) redox homeostasis | At delivery
  Redox homeostasis will be assessed in maternal blood using a biological assay to measure the capacity of the sample to prevent the oxidation of a known fluorescence probe, in the presence of an oxidant. The unit of measure is concentration of plasma expressed as equivalent to a know antioxidant (after performing a calibration curve).
Placental redox homeostasis | At delivery
  Redox homeostasis will be assessed in maternal blood using a biological assay to measure the capacity of the sample to prevent the oxidation of a known fluorescence probe, in the presence of an oxidant. The unit of measure is concentration of plasma expressed as equivalent to a know antioxidant (after performing a calibration curve).
Maternal inflammatory profile | between 24th and 28th gestational week
  Inflammatory profile will be assessed in maternal blood using a commercial kit to measure cytokines using ELISA assay, expressed as concentration per volume of sample.
Maternal inflammatory profile [change] | between 34th and 35th gestational week
  Inflammatory profile will be assessed in maternal blood using a commercial kit to measure cytokines using ELISA assay, expressed as concentration per volume of sample.
Fetal (cord blood) inflammatory profile | At delivery
  Inflammatory profile will be assessed in maternal blood using a commercial kit to measure cytokines using ELISA assay, expressed as concentration per volume of sample.
Placental inflammatory profile | At delivery
  Inflammatory profile will be assessed in maternal blood using a commercial kit to measure cytokines using ELISA assay, expressed as concentration per volume of sample.
Maternal metabolic profile | between 24th and 28th gestational week
  Metabolic profile will be assesses in maternal blood using Nuclear Magnetic Resonance metabolomics which measure small molecules (<1,500 Da) in the biological sample. The unit is intensity of the peak measured in a known volume/mass of sample obtained from the nuclear magnetic resonance spectra
Maternal metabolic profile [change] | between 34th and 35th gestational week
  Metabolic profile will be assesses in maternal blood using Nuclear Magnetic Resonance metabolomics which measure small molecules (<1,500 Da) in the biological sample. The unit is intensity of the peak measured in a known volume/mass of sample obtained from the nuclear magnetic resonance spectra
Fetal (cord blood) metabolic profile | At delivery
  Metabolic profile will be assesses in maternal blood using Nuclear Magnetic Resonance metabolomics which measure small molecules (<1,500 Da) in the biological sample. The unit is intensity of the peak measured in a known volume/mass of sample obtained from the nuclear magnetic resonance spectra
Placental metabolic profile | At delivery
  Metabolic profile will be assesses in maternal blood using Nuclear Magnetic Resonance metabolomics which measure small molecules (<1,500 Da) in the biological sample. The unit is intensity of the peak measured in a known volume/mass of sample obtained from the nuclear magnetic resonance spectra
Placental mitochondrial function at delivery | At delivery
  Mitochondrial function will be assessed using an electrode sensitive to oxygen which measures the decrease in oxygen tension in the chamber after addition of substrates and modulators of mitochondrial oxidative phosphorylation. This will be assessed in placental tissue and the units is concentration of oxygen per mass per time.

SECONDARY OUTCOMES:
Placental lipid metabolism | At delivery
  To investigate the alterations in lipid metabolism as a function of pre-gestational maternal obesity and gestational diabetes mellitus. Lipid metabolism will be assessed by lipid analysis using mass spectrometry to identify the major categories and lipid species in maternal, fetal and placental tissue. The unit is relative abundance per mass of tissue and volume of plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana El-Bacha, DSc, Principal Investigator — UFRJ; Carolina S Ferreira, DSc, Study Chair — UFRJ; Deborah AB Guimarães, DSc, Study Chair — UFRJ; Gabriela DA Pinto, DSc, Study Chair — UFRJ; Vanessa A Goes, DSc, Study Chair — UFRJ
Locations (1):
- Maternidade Escola da UFRJ, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It might be available if there is enough funding to perform RNA sequencing and DNA methylation in placental samples. The data to be shared will involved differential expressed genes and methylation sites in the placenta in order to help the investigation of the placental role in the origins of chronic diseases.